CLINICAL TRIAL: NCT01118546
Title: Physiopathology of Rapid Aspirin Desensitization in Patients With Coronary Artery Disease and a History of Hypersensitivity to Aspirin or NSAIDs
Brief Title: Physiopathology of Rapid Aspirin Desensitization
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P051026
Record Dates: First submitted 2010-03-31; First posted 2010-05-06 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2015-02

CONDITIONS: Hypersensitivity; Coronary Artery Disease
Keywords: aspirin; coronary artery disease; hypersensitivity; Platelet aggregation
MeSH Terms: conditions — Hypersensitivity; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- controls 2: patient without CAD, not on aspirin and without history of hypersensitivity
- case of hypersensitivity: patient with CAD on aspirin, with a history of hypersensitivity
- controls 1: patient with CAD on aspirin, without history of hypersensitivity

SUMMARY:
Aspirin is very effective in protecting patients with coronary artery disease against adverse cardiac events, because it is a potent "antiplatelet agent". Some patients may develop a history of hypersensitivity to aspirin and treatment cannot usually be resumed in these patients. We have developed a rapid procedure to induce tolerance in these patients (SILBERMAN et al, Am J CARDIOL 2005;95:509-10) and wish to test whether aspirin is as effective as antiplatelet agent in patients with a history of allergy to aspirin and who undergo desensitization as it is in patients without history of hypersensitivity

DETAILED DESCRIPTION:
Previous studies in allergology have proved the safety of desensitization procedures in allergic patients with an imperative indication for a medication. This tolerance state is usually obtained after a cumbersome procedure requiring several hours to days. We have adapted successfully such a procedure to the patients with acute coronary artery disease requiring urgent aspirin (excluding the ST elevation myocardial infarction) (SILBERMAN et al, Am J CARDIOL 2005;95:509-10).

Patients with a history of Aspirin or NonSteroidal Anti-Inflammatory Drugs hypersensitivity appear to have alterations of eicosanoid metabolism : these drugs trigger an imbalance toward the leucotriene pathway. This case-control study aims to

* evaluate after desensitization therapy the anti-aggregant effect of aspirin in these very particular patients : clinical outcome, PFA test, levels of the urinary metabolite of thromboxane A2 (11 dehydro thromboxane B2) and also usual aggregation tests.
* assess the in VITRO basophil activation induced by aspirin before and after desensitization procedure by flow cytometric cellular allergen test using basophils surface marker and mediators' dosage. Before the challenge procedure these tests aim to confirm the clinically established diagnosis of hypersensitivity. After desensitization, these tests intend to better assess the efficiency of the induced tolerance, to attempt to identify predictors of successful desensitization as well as identify potential cross reactivity with other NSAIDs..

This procedure is indicated in all patients with aspirin or NSAID intolerance with imperative cardiological indications for aspirin, such as acute coronary syndrome, or placement of a stent. The desensitization procedure must be performed in a coronary care unit; the patients are duly informed about benefits and risks of the challenge and provide written informed consent. Desensitization consists in rapidly escalating aspirin dose administration with ad hoc aspirin capsules prepared by the hospital pharmacist. Blood and urinary samples are obtained during the hospital stay for coronary and desensitization care. An additional blood and urine sample will be obtained 6 to 8 weeks later during an outpatient visit in the laboratory. Initial biological data will be compared to those of two control groups matched for age, gender and type of acute coronary syndrome :

* Controls 1: patients with CAD on aspirin, without history of hypersensitivity
* Controls 2: patients without CAD, not on aspirin and without history of hypersensitivity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age > 18 years
* Admitted to Hospital BICHAT, in Cardiology
* Patients with aspirin or NSAID intolerance due to hypersensitivity
* Imperative cardiological indications for aspirin, such as acute coronary syndrome, or placement of a stent
* Written informed consent
* Patient with health insurance coverage

EXCLUSION CRITERIA:

* Ongoing ST elevation acute coronary syndrome
* Ongoing signs or symptoms of hypersensitivity or allergy (asthma, urticaria, Quincke' edema, or other allergic symptoms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease and a history of aspirin hypersensitivity, requiring treatment with aspirin , referred to an academic tertiary center for desensitization
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2007-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation in response to arachidonic acid Basophil activation tests Platelet aggregation in response to arachidonic acid Basophil activation tests | day 1, after aspirin desensitization

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel STEG, Pr, Principal Investigator — APHP
Locations (1):
- Centre hospitalier Bichat Claude Bernard, Paris, France

REFERENCES:
- See also: Publication — http://www.ncbi.nlm.nih.gov/pubmed/27533953